CLINICAL TRIAL: NCT04000087
Title: Electrocardiogram Artificial Intelligence-Guided Screening for Low Ejection Fraction (EAGLE)
Brief Title: ECG AI-Guided Screening for Low Ejection Fraction
Acronym: EAGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiaoxi Yao, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-003137
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Asymptomatic Left Ventricular Systolic Dysfunction (Disorder); Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Care teams randomized to intervention will have access to the screening tool.
  Interventions: Other: AI-enabled ECG-based Screening Tool
- Control (No Intervention): Care teams randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool — A novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis and management of left ventricular systolic dysfunction.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial (RCT) to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis and management of left ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinicians who are part of a participating care team that care for adult patients and have the ability to order ECG and TTE (this includes physicians, nurse practitioners, and physician assistants).

Exclusion Criteria:

* Primary care clinicians working in pediatrics, acute care, nursing homes, and resident care teams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
New Diagnosis of Low Ejection Fraction (defined as ejection fraction ≤50%) | Within 90 days
  Ejection fraction obtained by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Yao, PhD, MPH, Principal Investigator — Mayo Clinic; Peter Noseworthy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Yao X, McCoy RG, Friedman PA, Shah ND, Barry BA, Behnken EM, Inselman JW, Attia ZI, Noseworthy PA. ECG AI-Guided Screening for Low Ejection Fraction (EAGLE): Rationale and design of a pragmatic cluster randomized trial. Am Heart J. 2020 Jan;219:31-36. doi: 10.1016/j.ahj.2019.10.007. Epub 2019 Oct 25. PMID 31710842
- [Derived] Barry B, Zhu X, Behnken E, Inselman J, Schaepe K, McCoy R, Rushlow D, Noseworthy P, Richardson J, Curtis S, Sharp R, Misra A, Akfaly A, Molling P, Bernard M, Yao X. Provider Perspectives on Artificial Intelligence-Guided Screening for Low Ejection Fraction in Primary Care: Qualitative Study. JMIR AI. 2022 Oct 14;1(1):e41940. doi: 10.2196/41940. PMID 38875550
- [Derived] Zahrieh D, Croghan IT, Inselman JW, Mandrekar SJ. Guidelines for Data and Safety Monitoring in Pragmatic Randomized Clinical Trials Using Case Studies. Mayo Clin Proc. 2023 Nov;98(11):1712-1726. doi: 10.1016/j.mayocp.2023.02.019. PMID 37923529
- [Derived] Rushlow DR, Croghan IT, Inselman JW, Thacher TD, Friedman PA, Yao X, Pellikka PA, Lopez-Jimenez F, Bernard ME, Barry BA, Attia IZ, Misra A, Foss RM, Molling PE, Rosas SL, Noseworthy PA. Clinician Adoption of an Artificial Intelligence Algorithm to Detect Left Ventricular Systolic Dysfunction in Primary Care. Mayo Clin Proc. 2022 Nov;97(11):2076-2085. doi: 10.1016/j.mayocp.2022.04.008. PMID 36333015
- [Derived] Yao X, Rushlow DR, Inselman JW, McCoy RG, Thacher TD, Behnken EM, Bernard ME, Rosas SL, Akfaly A, Misra A, Molling PE, Krien JS, Foss RM, Barry BA, Siontis KC, Kapa S, Pellikka PA, Lopez-Jimenez F, Attia ZI, Shah ND, Friedman PA, Noseworthy PA. Artificial intelligence-enabled electrocardiograms for identification of patients with low ejection fraction: a pragmatic, randomized clinical trial. Nat Med. 2021 May;27(5):815-819. doi: 10.1038/s41591-021-01335-4. Epub 2021 May 6. PMID 33958795
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials